CLINICAL TRIAL: NCT01132755
Title: Rapid Gastric and Pancreas Cancer Staging Utilizing Peritoneal Lavage
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10-011
Record Dates: First submitted 2010-05-26; First posted 2010-05-28 (Estimated); Results first posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2017-08

CONDITIONS: Gastric Cancer; Pancreatic Cancer
Keywords: gastric; pancreas; laparoscopy; peritoneal lavage; 10-011; gastric and pancreatic cancer
MeSH Terms: conditions — Stomach Neoplasms; Pancreatic Neoplasms | interventions — Peritoneal Lavage; Therapeutic Irrigation; Fluid Therapy

ARMS (1):
- Patients who require diagnostic laparoscopy (Experimental): Diagnostic peritoneal lavage will be performed at the time of laparoscopy utilizing a Veress needle/Seldinger technique to insert a peritoneal dialysis catheter. This is not a new technique. The Veress needle will be inserted in the abdominal wall, at a site to be left up to the individual surgeon.
  Interventions: Procedure: Diagnostic peritoneal lavage

INTERVENTIONS:
Procedure: Diagnostic peritoneal lavage — The Veress needle will be inserted in the abdominal wall, at a site to be left up to the individual surgeon. Caudal traction will be applied to the abdominal wall to provide a firm abdominal wall to insert the needle through, minimizing the peritoneum from tenting down closer to visceral structures. Intraperitoneal placement of the catheter will be confirmed by injection of saline into the needle with no resistance and with the saline in the hub of the needle falling into the peritoneal cavity spontaneously. A guide wire will be placed through the Veress and utilizing the Seldinger technique, a 9Fr peritoneal catheter will be placed.
  Other Names: 800cc of saline will be infused and 60ml will be extracted and sent to the; cytopathology lab. When the laparoscope is inserted for laparoscopic guided; lavage, no additional fluid will be instilled, unless there is no available; fluid in the RUQ, LUQ, and pelvic locations that are currently sampled.; Instead, the fluid already present from the percutaneous lavage will be; utilized.

SUMMARY:
This study is being done to develop a new method that can rapidly stage patients with gastric and pancreas cancer. Staging means finding out what is the extent of the cancer in a patient's body.

Currently before patients have the surgery to remove their cancer, a surgical exam is done in the operating room to see if their cancer has spread. A thin tube-like instrument with lens and a light is placed into the abdomen. This is done by making small cuts into the body. This exam is called a diagnostic laparoscopy. If cancer spread is not seen, fluid is put into the abdomen and then taken out. This is called "lavage" or washing. The fluid is then looked at in a laboratory. If the fluid contains cancer cells surgery is often delayed.

The investigators are testing a new method to put the fluid into the abdomen. It is called percutaneous lavage. Percutaneous means "through the skin". A needle is put through the skin into the abdomen. Tubing is then placed over the needle so that fluid can be put into the abdomen and then taken out. The fluid is then looked at in a laboratory. The investigators want to see if the two methods are equal because if they are equal, in the future, patients may be able to have this procedure done outside of the operating room.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 years of age and older
* Informed consent in keeping with the policies of Memorial Sloan-Kettering Cancer Center
* Presentation of gastric or pancreatic cancer based on objective findings by either:

  * CT scan
  * Endoscopy
  * Pathologic examination
* Candidate for surgical treatment and are scheduled for laparoscopy with peritoneal lavage.

Exclusion Criteria:

* Under 18 years of age
* Inability to speak or read English, and an appropriate translator is not identifiable
* Unable or unwilling to give informed consent
* Patients with synchronous cancers of other abdominal organs
* Multiple prior surgical procedures on the abdomen where the surgeon feels that percutaneous lavage may be dangerous.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2017-08-16 (Actual); Study Completion 2017-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: T. Peter Kingham, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients Who Require Diagnostic Laparoscopy
Started | 112
Completed | 70
Not Completed | 42
Not completed — Procedure not done due to medical reason | 23
Not completed — Protocol Violation | 15
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Patients Who Require Diagnostic Laparoscopy
Number analyzed (Participants) | 112
Age, Continuous [Median (Full Range); unit: years] | 65 [38 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 106
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 87
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 112

OUTCOME MEASURES:

1. Primary Outcome: Number of Study Participants With Adequate Percutaneous Lavage Specimen Collection
Description: Cytology will be performed to compare percutaneous and laparoscopic lavage results in order to determine if percutaneous lavage specimen collection is concordant with laparoscopic lavage results
Time Frame: 2 years
Population: 76 participants underwent percutaneous and laparoscopic lavage
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Who Require Diagnostic Laparoscopy
Number analyzed (Participants) | 76
Participants
  Percutaneous & laparoscopic specimen collection | 70
  Inability to access abdomen using Veress needle | 2
  Inadequate fluid return for cytology | 4

2. Secondary Outcome: Safety of Peritoneal Lavage in Place of Laparoscopic Lavage.
Description: Safety is measured in the number of bowel, major omental, or major vascular injuries.
Time Frame: 2 years
Measure: Number; unit: procedural injuries
Arm/Group | Patients Who Require Diagnostic Laparoscopy
Number analyzed (Participants) | 76
procedural injuries | 0

ADVERSE EVENTS:
Time Frame: Up to 83 Months
Arm/Group | Patients Who Require Diagnostic Laparoscopy
All-Cause Mortality (participants affected / at risk) | 73/115
Serious Adverse Events (participants affected / at risk) | 0/115
Other Adverse Events (participants affected / at risk) | 0/115

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-19): https://cdn.clinicaltrials.gov/large-docs/55/NCT01132755/Prot_SAP_000.pdf